CLINICAL TRIAL: NCT02399449
Title: Evaluation of Iron Species in Healthy Subjects Treated With Generic and Reference Sodium Ferric Gluconate
Brief Title: IV Iron Safety: Evaluation of Iron Species in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, James E Polli, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00060573
Record Dates: First submitted 2015-03-02; First posted 2015-03-26 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Anemia
Keywords: iron; pharmacokinetics
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brand sodium ferric gluconate then Generic sodium ferric gluconate (Experimental): Crossover trial. Each arm will receive Brand sodium ferric gluconate (single dose of 125mg) then Generic sodium ferric gluconate (single dose of 125mg)
  Interventions: Drug: Brand sodium ferric gluconate; Drug: Generic sodium ferric gluconate
- Generic sodium ferric gluconate then Brand sodium ferric gluconate (Experimental): Crossover trial. Each arm will receive Generic sodium ferric gluconate (single dose of 125mg) then Brand sodium ferric gluconate (single dose of 125mg)
  Interventions: Drug: Brand sodium ferric gluconate; Drug: Generic sodium ferric gluconate

INTERVENTIONS:
Drug: Brand sodium ferric gluconate — brand product
  Other Names: Ferrecit
Drug: Generic sodium ferric gluconate — generic product
  Other Names: generic iron

SUMMARY:
An approved treatment for anemia or low blood count due to chronic kidney disease is IV (intravenous, given into the vein) injection of an iron treatment. IV iron increases iron in the blood. Many IV iron therapies are now available in both brand name and generic forms. One common IV iron product is sodium ferric gluconate (SFG) sold as brand name Ferrlecit. Recently, a generic version of Ferrlecit was approved but was felt to be possibly more toxic than the brand product. The purpose of this research project is to see if the brand and generic IV iron products produce the same amount of iron in the blood in healthy volunteers, including an iron form that more toxic than other iron forms.

DETAILED DESCRIPTION:
A generic version of Ferrlecit was approved in 2011 and is available. Shortly after the approval of the generic, a 'Reflections Paper on Non-Clinical Studies for Generic Nanoparticle Iron Medicinal Product Applications' was published by the European Medicines Agency. The authors of this paper proposed that generic iron preparations deliver increased levels of 'labile iron' to the plasma resulting in oxidative damage and toxicity. As such, studies measuring the in vivo levels of free or labile iron from generic versus brand iron-preparations were recommended.

The primary outcome will be the assessment of non-inferiority of the generic colloid product against the reference colloid product with respect to non-transferrin bound iron (NTBI), after single-dose i.v. administration of brand and generic sodium ferric gluconate injections in n=48 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* View 1 Males or female, with age 18-65 years old, systolic blood pressure within 90-150, and diastolic blood pressure within 60-90
* View 2 Healthy volunteers: Subjects in good health including being iron replete and not anemic, as determined by screening evaluation that is not greater than 30 days before the first drug study visit
* View 3 Willing to avoid caffeine containing products 24 hours prior to and day of study visits
* View 4 Willing to stop all OTC medications for 24 hours prior to and during study visits
* View 5 Able to provide informed consent

Exclusion Criteria:

* View 1 Presence of significant medical disease (including cardiovascular, pulmonary, hematologic, endocrine, immunologic, neurologic, gastrointestinal or psychiatric)
* View 2 Subjects who are iron deficient or with iron overload
* View 3 Presence of hepatic or renal disease
* View 4 Pregnant women, breast feeding or trying to become pregnant
* View 5 Excessive alcohol use (i.e. current physical, behavioral, or personal manifestations related to the abuse or dependency on alcohol)
* View 6 Routine use (i.e. daily or weekly) prescription medication except birth control pills
* View 7 Currently taking iron in any form (e.g. oral or IV)
* View 8 Allergic to IV iron, including sodium ferric gluconate, or any of its inactive components, including benzyl alcohol
* View 9 Undergoing therapy for solid tumor or blood malignancy
* View 10 Any condition in which in the opinion of the PI or medical physician would increase risk to the subject or interfere with the integrity of the study
* View 11 Donated blood within last 56 days of screening. Received IV iron or RBC transfusion(s) 10 days prior to screening. Plan to donate blood, or receive IV iron or RBC transfusion(s), during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Polli, Principal Investigator — U of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

REFERENCES:
- [Background] Baribeault D. Sodium ferric gluconate (SFG) in complex with sucrose for IV infusion: bioequivalence of a new generic product with the branded product in healthy volunteers. Curr Med Res Opin. 2011 Aug;27(8):1653-7. doi: 10.1185/03007995.2011.597738. Epub 2011 Jun 30. PMID 21714710

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment number is the number of participants who signed a consent form, per local IRB requirements.
Groups:
- Brand Sodium Ferric Gluconate Then Generic Sodium Ferric Gluconate: Crossover trial. Each arm will receive Brand sodium ferric gluconate then Generic sodium ferric gluconate
  Brand sodium ferric gluconate: brand product
  Generic sodium ferric gluconate: generic product
- Generic Sodium Ferric Gluconate Then Brand Sodium Ferric Gluconate: Crossover trial. Each arm will receive Generic sodium ferric gluconate then Brand sodium ferric gluconate
  Brand sodium ferric gluconate: brand product
  Generic sodium ferric gluconate: generic product
Period: Overall Study
Arm/Group | Brand Sodium Ferric Gluconate Then Generic Sodium Ferric Gluconate | Generic Sodium Ferric Gluconate Then Brand Sodium Ferric Gluconate
Started | 25 | 32
Completed | 22 | 22
Not Completed | 3 | 10
Not completed — Withdrawal by Subject | 3 | 9
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brand Sodium Ferric Gluconate Then Generic Sodium Ferric Gluconate | Generic Sodium Ferric Gluconate Then Brand Sodium Ferric Gluconate | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 34 [22 to 56] | 36 [22 to 54] | 35 [22 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 7 | 12 | 19
  More than one race | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Non-transferrin Bound Iron
Description: area under curve of non-transferrin bound iron. Non-transferrin bound iron is the difference between plasma total iron and transferrin bound iron, both of which were directly quantified. Units are concentration x time (i.e. ppb x hr).
Time Frame: 0-36 hr
Measure: Mean (Standard Error); unit: ppb x hours
Arm/Group | Brand Sodium Ferric Gluconate | Generic Sodium Ferric Gluconate
Number analyzed (Participants) | 35 | 35
ppb x hours | 56230 (2910) | 61250 (3410)

2. Secondary Outcome: Plasma Total Iron
Description: area under curve of plasma total iron. Units are concentration x time (i.e. ppb x hr).
Time Frame: 0-36 hr
Measure: Mean (Standard Error); unit: ppb x hours
Arm/Group | Brand Sodium Ferric Gluconate | Generic Sodium Ferric Gluconate
Number analyzed (Participants) | 35 | 35
ppb x hours | 132800 (4700) | 134700 (5100)

3. Secondary Outcome: Transferrin Bound Iron
Description: area under curve of transferrin bound iron. Units are concentration x time (i.e. ppb x hr).
Time Frame: 0-36 hr
Measure: Mean (Standard Error); unit: ppb x hours
Arm/Group | Brand Sodium Ferric Gluconate | Generic Sodium Ferric Gluconate
Number analyzed (Participants) | 35 | 35
ppb x hours | 96760 (3680) | 91740 (3980)

ADVERSE EVENTS:
Time Frame: About 1 month
Arm/Group | Brand Sodium Ferric Gluconate | Generic Sodium Ferric Gluconate
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/46
Other Adverse Events (participants affected / at risk) | 13/47 | 3/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brand Sodium Ferric Gluconate (N=47) | Generic Sodium Ferric Gluconate (N=46)
hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brand Sodium Ferric Gluconate (N=47) | Generic Sodium Ferric Gluconate (N=46)
Abdominal Cramping (General disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Leg Swelling (General disorders) | 1 (1) | 0 (0)
Lower Back Pain (General disorders) | 7 (7) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Infusion Site Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Facial Flushing (General disorders) | 1 (1) | 0 (0)
Infusion Site Pain (General disorders) | 0 (0) | 1 (1)
Infusion Site-To -Hand Swelling (General disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Finger Cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 0 (0)
Hand Swelling (General disorders) | 2 (2) | 0 (0)
Hand Muscle Stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT02399449/Prot_SAP_001.pdf